CLINICAL TRIAL: NCT04720443
Title: A Phase 1, Two-Part Study of NIP292 Tablets in Healthy Adult Subjects: Part 1 - Randomized, Double-Blind, Placebo-Controlled Assessment of Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses; Part 2 - Randomized, Double-Blind, Placebo-Controlled Assessment of Safety, Tolerability and Pharmacokinetics of Multiple Ascending Oral Doses.
Brief Title: A Safety, Tolerability, and Pharmacokinetic Study of NIP292 in Healthy Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The National Institutes of Pharmaceutical R&D Co. Ltd, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NIP292-101
Record Dates: First submitted 2020-12-30; First posted 2021-01-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SAD Part 1 Cohort 1 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet at 10 mg) or placebo. In each cohort, to mitigate any unforeseen safety issues, the first 2 subjects (1 active + 1 placebo) will be admitted and dosed, and at least 48 hours apart from the other 6 subjects. The remaining 6 subjects of each cohort will be dosed after review of the safety data of the first 2 subjects.
  Interventions: Drug: NIP292 tablet
- SAD Part 1 Cohort 2 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet at 30 mg) or placebo. In each cohort, to mitigate any unforeseen safety issues, the first 2 subjects (1 active + 1 placebo) will be admitted and dosed, and at least 48 hours apart from the other 6 subjects. The remaining 6 subjects of each cohort will be dosed after review of the safety data of the first 2 subjects.
  Interventions: Drug: NIP292 tablet
- SAD Part 1 Cohort 3 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet at 100mg) or placebo. In each cohort, to mitigate any unforeseen safety issues, the first 2 subjects (1 active + 1 placebo) will be admitted and dosed, and at least 48 hours apart from the other 6 subjects. The remaining 6 subjects of each cohort will be dosed after review of the safety data of the first 2 subjects.
  Interventions: Drug: NIP292 tablet
- SAD Part 1 Cohort 4 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet at 300 mg) or placebo. In each cohort, to mitigate any unforeseen safety issues, the first 2 subjects (1 active + 1 placebo) will be admitted and dosed, and at least 48 hours apart from the other 6 subjects. The remaining 6 subjects of each cohort will be dosed after review of the safety data of the first 2 subjects.
  Interventions: Drug: NIP292 tablet
- SAD Part 1 Cohort 5 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet at 500 mg)or placebo. In each cohort, to mitigate any unforeseen safety issues, the first 2 subjects (1 active + 1 placebo) will be admitted and dosed, and at least 48 hours apart from the other 6 subjects. The remaining 6 subjects of each cohort will be dosed after review of the safety data of the first 2 subjects.
  Interventions: Drug: NIP292 tablet
- MAD Part 2 Cohort 1 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet dosage 1) or placebo. All subjects will receive either NIP292 or placebo on an empty stomach for 7 days (from Day 1 to Day 7), and dosing frequency will be identical and either QD, Q12H, or Q8H (depending on the observed PK data in Part 1). Two dose levels (dose 1 and dose 2) proposed for MAD part will be determined based on the doses evaluated in SAD part.
  Interventions: Drug: NIP292 tablets
- MAD Part 2 Cohort 2 (Experimental): Eight subjects will be randomized at a ratio of 3:1 in each cohort to receive either NIP292 (oral tablet dosage 2) or placebo. All subjects will receive either NIP292 or placebo on an empty stomach for 7 days (from Day 1 to Day 7), and dosing frequency will be identical and either QD, Q12H, or Q8H (depending on the observed PK data in Part 1). Two dose levels (dose 1 and dose 2) proposed for MAD part will be determined based on the doses evaluated in SAD part.
  Interventions: Drug: NIP292 tablets

INTERVENTIONS:
Drug: NIP292 tablet — NIP292 (oral tablet at 10 mg) or placebo
  Arms: SAD Part 1 Cohort 1
Drug: NIP292 tablet — NIP292 (oral tablet at 30 mg) or placebo
  Arms: SAD Part 1 Cohort 2
Drug: NIP292 tablet — NIP292 (oral tablet at 100 mg) or placebo
  Arms: SAD Part 1 Cohort 3
Drug: NIP292 tablet — NIP292 (oral tablet at 300 mg) or placebo
  Arms: SAD Part 1 Cohort 4
Drug: NIP292 tablet — NIP292 (oral tablet at 500 mg) or placebo
  Arms: SAD Part 1 Cohort 5
Drug: NIP292 tablets — NIP292 (oral tablet at dosage 1) or placebo
  Arms: MAD Part 2 Cohort 1
Drug: NIP292 tablets — NIP292 (oral tablet at dosage 2) or placebo
  Arms: MAD Part 2 Cohort 2

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of single ascending and multiple ascending oral doses of NIP292 tablets administered following an overnight fast in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (non-childbearing potential) subjects between age 18 and 55 years (inclusive), in general good health without clinically significant abnormalities.
2. Female subjects of non-childbearing potential will be authorized to participate in this study if at least one of the following criteria are met:

   1. Surgical sterilization (e.g., hysterectomy, bilateral oophorectomy and/or bilateral salpingectomy, but excluding bilateral tubal occlusion);
   2. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state (with a single repeat permitted if deemed necessary by the investigator); and β-human chorionic gonadotropin (β-HCG) is negative at screening and the admission.
3. Body mass index (BMI) of 18-32 kg/m2 (inclusive), and a total body weight >50 kg (110 lb).
4. Clinical laboratory values within the normal limits as defined by the clinical laboratory. Of note, individual values out of normal range can be accepted if judged as not clinically significant by the investigator. Repeat assessment can be conducted at the discretion of the investigator or delegate.
5. Subjects who are willing and able to comply with the prescribed protocol treatment and evaluations.
6. Subjects must provide signed written informed consent prior to any study-specific procedures.

Exclusion Criteria:

Subjects with any of the following characteristics or conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies).
2. History of drug abuse in the past 5 years, or a positive urine drug test at screening or the admission.
3. History of excessive alcohol intake exceeding 14 drinks/week (1 drink = 5 ounces [150 mL] of wine, or 12 ounces [360 mL] of beer, or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening, or a positive alcohol breath test at screening or the admission.
4. Current smoker, or difficulty abstaining from smoking for the duration of study confinement.
5. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
6. Use of prescription or nonprescription drugs or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication; however, limited use of nonprescription medications that are not believed to affect the overall results of the study may be permitted on a case by case basis following approval by the investigator and the Sponsor.
7. Previous participation in this study; subjects can only be randomized and receive the study medication in 1 of the 2 parts in this study.
8. Any condition possibly affecting drug absorption per the principal investigator's discretion (e.g., gastrectomy).
9. Screening supine systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg. If SBP ≥140 mmHg or DBP ≥90 mmHg, the blood pressure assessment should be repeated 2 more times and the average of the 3 blood pressure values should be used to determine the subject's eligibility.
10. Screening supine 12-lead ECG demonstrating a QTcF (using Fridericia's formula, QTcF = QT/RR1/3) interval >450 msec for males or >470 msec for females,or a QRS interval >120 msec. If QTcF >450 msec or QRS >120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the subject's eligibility.
11. Subjects with history of hepatitis, or positive result at screening for hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), hepatitis C antibody (HCVAb), or human immunodeficiency virus antibody (HIVAb).
12. Pregnant female subjects; breastfeeding female subjects; male subjects able to father children who are unable to use a highly effective method of contraception for the duration of the study and for at least 90 days after the last dose of study medication.
13. Blood donation (excluding plasma donations) of approximately 450 mL or more within 60 days prior to the first dose of study medication.
14. History of sensitivity to heparin or heparin induced thrombocytopenia (if heparin is used to flush intravenous catheters used during serial blood collections).
15. Unwilling or unable to comply with this study protocol.
16. Any other medical or psychiatric condition that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence, potential significance, and clinical importance of adverse events (AE) after single dose of NIP292 in 48 healthy subject. | 31 days
  The AEs developed during or after the study treatment (as treatment-emergent adverse event [TEAE]) will be summarized by preferred term, system organ class, severity, and relationship to the investigational product.
To evaluate the incidence, potential significance, and clinical importance of adverse events (AE) after multipe dose of NIP292 in 24 healthy subject. | 37 days
  The AEs developed during or after the study treatment (as treatment-emergent adverse event [TEAE]) will be summarized by preferred term, system organ class, severity, and relationship to the investigational product.
The change of Clinical Laboratory Tests | 31 days in SAD
  Descriptive statistics of absolute values and changes from baseline will be summarized by dose/regimen and time. Laboratory abnormalities will be tabulated by time.
The change of Clinical Laboratory Tests | 37 days in MAD
  Descriptive statistics of absolute values and changes from baseline will be summarized by dose/regimen and time. Laboratory abnormalities will be tabulated by time.
Electrocardiogram (ECG) | 31 days in SAD
  Changes from baseline for the ECG parameters (i.e., QT, heart rate, QTcF, PR and QRS) will be summarized by dose/regimen and time. The number (%) of subjects with maximum post-dose QTcF values and maximum increases from baseline will be tabulated by regimen.
Electrocardiogram (ECG) | 37 days in MAD
  Changes from baseline for the ECG parameters (i.e., QT, heart rate, QTcF, PR and QRS) will be summarized by dose/regimen and time. The number (%) of subjects with maximum post-dose QTcF values and maximum increases from baseline will be tabulated by regimen.

SECONDARY OUTCOMES:
To characterize the maximum plasma concentration(Cmax) of NIP292 tablets in 48 healthy adult subjects. | 31 days
  PK parameters derived from plasma NIP292 concentration data following single oral doses: maximum plasma concentration(Cmax)
To characterize the time to maximum plasma concentration (Tmax) of NIP292 tablets in 48 healthy adult subjects. | 31 days
  PK parameters derived from plasma NIP292 concentration data following single oral doses: time to maximum plasma concentration (Tmax)
To characterize the time to area under the concentration-time curve from hour 0 to last postdose(AUC0-last) of NIP292 tablets in 48 healthy adult subjects. | 31 days
  PK parameters derived from plasma NIP292 concentration data following single oral doses: area under the concentration-time curve from hour 0 to last postdose(AUC0-last)
To characterize the maximum plasma concentration(Cmax) of NIP292 tablets in 24 healthy adult subjects. | 37 days
  PK parameters derived from plasma NIP292 concentration data following multiple oral doses: maximum plasma concentration (Cmax)
To characterize the time to maximum plasma concentration (Tmax) of NIP292 tablets in 24 healthy adult subjects. | 37 days
  PK parameters derived from plasma NIP292 concentration data following multiple oral doses: time to maximum plasma concentration (Tmax)
To characterize the area under the concentration-time curve from hour 0 to last postdose(AUC0-last) of NIP292 tablets in 24 healthy adult subjects. | 37 days
  PK parameters derived from plasma NIP292 concentration data following multiple oral doses:area under the concentration-time curve from hour 0 to last postdose(AUC0-last)
To characterize the renal clearance of NIP292 tablets, if data permit | 37 days
  the urine PK parameters:renal clearance(CLr)

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL International, Glendale, California, United States